CLINICAL TRIAL: NCT01780415
Title: Genomic DNA in Human Blastocoele Fluid
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cervesi Hospital, Cattolica, Italy (Other)
Responsible Party: Principal Investigator, Palini Simone, Senior Clinical Embryologist, Cervesi Hospital, Cattolica, Italy
Other Study IDs: NewEra21972
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Chromosomal Aneuploidies; Single Gene Desease
Keywords: Blastocoele fluid; Human DNA; molecular diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bastovit: all the patients that have supernumerary embryos to vitrify at blastocyst stage
  Interventions: Other: blastocoele aspiration

INTERVENTIONS:
Other: blastocoele aspiration

SUMMARY:
The objective will focus on the characterization of DNA fragments present in Blastocoele fluid, and the evaluation of these fragments as potential target for Preimplantation Genetic Diagnosis. To reach this goal, real-time PCR, Whole Genome Amplification techniques and -subsequently- Next Generation Sequencing and aCGH approaches will be used.

ELIGIBILITY:
Inclusion Criteria:

* IVF patient with supernumerary embryos to vitrify at blastocyst stage

Exclusion Criteria:

* IVF patient without blastocyst formation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: IVF patient with supernumerary embryos to vitrify at blastocyst stage
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Number of samples with DNA in blastocoele Fluid | 6 month
  the presence of DNA will be evaluated through rtPCR

SECONDARY OUTCOMES:
Number of euploid samples | 8 months
  Array CGH

CONTACTS AND LOCATIONS:
Locations (1):
- Cervesi Hospital IVF Unit, Cattolica, Rimini, Italy